CLINICAL TRIAL: NCT00205062
Title: Pilot Study of the Role of PET-CT for Diagnosis and Assessment of Therapeutic Efficacy in Inflammatory Bowel Disease
Brief Title: Positron Emission Tomography (PET)-Computed Tomography (CT) in Inflammatory Bowel Disease (IBD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: No Accrual
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: M-2004-0251
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2008-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

INTERVENTIONS:
Procedure: PET-CT

SUMMARY:
The main hypothesis is that PET-CT will be a valuable diagnostic tool in diagnosing and evaluating treatment for IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patient with either Crohn's disease or ulcerative colitis whose disease is flaring

Exclusion Criteria:

* Indeterminate diagnosis, pregnant, breastfeeding, or other contraindication to PET-CT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Does this technique provide an accurate assessment of disease inflammation compared to standard clinical markers?

SECONDARY OUTCOMES:
Does this technique provide additional information for practitioners on extent of disease?

CONTACTS AND LOCATIONS:
Overall Officials: Randall Meisner, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States